CLINICAL TRIAL: NCT00568308
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Parallel-group, International, Multicentre Phase III Trial of PI-88 in the Adjuvant Treatment of Post-resection Hepatocellular Carcinoma
Brief Title: Phase III Study of PI-88 in Post-resection Hepatocellular Carcinoma
Acronym: PATHWAY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Commercial decision to discontinue the study
Sponsor: Progen Pharmaceuticals (Industry)
Responsible Party: Liz Wilson, Progen Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR88302
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Cancer; Liver Cancer; Primary Liver Cancer; Hepatocellular Carcinoma; Hepatoma
Keywords: Hepatocellular Carcinoma; PI-88; Phase III; Adjuvant Therapy; Hepatoma; Liver Cancer
MeSH Terms: conditions — Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — phosphomannopentaose sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: PI-88

INTERVENTIONS:
Drug: PI-88 — 160mg subcutaneous injection
  Arms: 2
Drug: placebo — matched placebo
  Arms: 1

SUMMARY:
The purpose of this study is to determine if PI-88 is effective and safe in patients who have had surgery to remove primary liver cancer.

DETAILED DESCRIPTION:
Primary liver cancer (hepatocellular carcinoma or HCC) is the fifth most common cancer worldwide. Surgery to remove the tumour remains the principal form of treatment for liver cancer, however recurrence of the disease after surgery is common and survival after recurrence is poor. At the moment there is no recommended standard treatment for HCC immediately after the tumour has been removed surgically. PI-88 is a new experimental drug which blocks the growth of new blood vessels in tumours to stop the tumour growing (starves it of food) and also stops tumour cells spreading. Previous experience with PI-88 has shown it has been well tolerated and has shown some benefit in delaying the time it takes for the hepatocellular carcinoma to reappear after surgery. The purpose of this study is to determine if PI-88 is effective and safe in patients who have had surgery to remove primary liver cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically-proven primary hepatocellular carcinoma with curative resection performed in the 4 - 6 weeks prior to randomisation.
* ECOG performance status 0 to 2
* Child Pugh classification A or B

Key Exclusion Criteria:

* Any evidence of tumour metastasis or co-existing malignant disease
* Any prior recurrence of HCC or any liver resection prior to the most recent procedure
* History of prior HCC therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Disease-free Survival | End of Study

SECONDARY OUTCOMES:
Overall Survival | End of study
Time to Recurrence | End of Study
Quality of Life | End of Study
Safety and Tolerability | End of Study
Compliance | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie TP Poon, MD, Principal Investigator — University of Hong Kong, Queen Mary Hospital
Locations (10):
- United States of America, New York, United States
- Australia, Australia
- Canada, Canada
- Hong Kong, Hong Kong
- Italy, Italy
- Malaysia, Malaysia
- Singapore, Singapore
- Spain, Spain
- Dawan, Taiwan
- Thailand, Thailand

REFERENCES:
- See also: Progen Pharmaceuticals Website — http://www.progen-pharma.com